CLINICAL TRIAL: NCT03486483
Title: The Slackline as a Rehabilitation Tool for Children and Teenagers With Spastic Cerebral Palsy: a Randomised Clinical Trial
Brief Title: Spastic Cerebral Palsy and Slackline
Acronym: SCPSLACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Santos (Other)
Responsible Party: Sponsor-Investigator, Luis Santos, Sponsor-Investigator, University of Oviedo
Organization: University of Oviedo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No. 53/2014
Record Dates: First submitted 2018-03-18; First posted 2018-04-03 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Slackline Training (Experimental): Supervised Slackline training in children and teenagers with spastic cerebral palsy (grade I and II of the Gross Motor Function Classification System). Intervention included 18 slackline rehabilitation sessions for 6 weeks: 3 sessions per week on non-consecutive days, 30 min each one.
  Interventions: Other: Exercise
- Physical Activity (No Intervention): The control group followed its usual weekly physical activity routine.

INTERVENTIONS:
Other: Exercise — Intervention included 18 slackline rehabilitation sessions for 6 weeks: 3 sessions per week on non-consecutive days, 30 min each one.
  Arms: Supervised Slackline Training

SUMMARY:
The aim of the present study was to assess whether supervised slackline training improves postural control in children and teenagers with spastic cerebral palsy (grade I and II of the Gross Motor Function Classification System).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with any expression of spastic cerebral palsy and rated I-II on the Gross Motor Functional classification.
* Between 9 and 16 years of age.
* Ability to cooperate with simple instructions.
* Able to stand for at least 2 min without assistance.
* Able to walk at least 10 m without assistance.

Exclusion Criteria:

* Individuals were excluded if they underwent neuro or orto surgery during or up to one year prior to the study, botulinum toxin injection or intrathecal pump during or up to six months prior to the study and/or rotational osteotomies, if they expressed gait deviations limited by musculoskeletal contracture, presented specific medical or orthopedic conditions that precluded exercising
* or if they did not meet the eligibility criteria.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Static posturography (a composite measure). | 6 weeks.
  The centre of pressure (CoP) parameters (these CoP parameters; Length, Xmean, Ymean, Xdeviation and Ydeviation in mm, Area in mm2 and Speed, Xspeed and Yspeed in m/s will be combined to report the static posturography).

SECONDARY OUTCOMES:
Myoelectrical activity. | 6 weeks.
  Soles, Tibialis Anterior and Peroneus Longus (myoelectrical activity in microvolts).
Jump Performance | 6 weeks.
  Countermovement Jump Test and Abalakov´s Test (jump height in cm).